CLINICAL TRIAL: NCT05161884
Title: Validation of a Non-invasive Assessment of Central Venous Oxygen Saturation by Using Magnetic Resonance Imaging
Brief Title: Validation of a Non-invasive Assessment of Central Venous Oxygen Saturation by Using MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: German Heart Institute (Other)
Responsible Party: Principal Investigator, Sebastian Kelle, Head of Cardiac MRI, German Heart Institute
Other Study IDs: EA4/118/20
Record Dates: First submitted 2021-11-16; First posted 2021-12-17 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Preclinical Study group: n=10 Landrace pigs The aim of the pre-clinical study was to assess the accuracy of BOLD-T2 MRI in acute systemic hyper- and hypoxemia in a porcine model in contrast to cardiac catheterization.
- Validation Study group: n=25 The patients have an indication for a right heart catheter examination. This is a routine diagnostic examination that is performed on these patients.
  Compared to the clinical routine, an additional MRI measurement will be performed. The measurement will be performed before the cardiac catheterization.
  For the MRI examination, the patient/subject is placed in a magnetic resonance imaging machine. The MRI examination initially includes approximately 15 minutes of standard images for orientation and determination of function, morphology, and tissue characteristics. This is followed by images to determine oxygen saturation in the ventricles (approximately 5 minutes).
  If a CMR examination is already planned for a patient for other reasons, this will only be extended by the recordings for the determination of oxygen saturation (approx. 5 minutes) at the time of study inclusion.
  During the MRI measurements, patients will also perform a stepper stress test.
- Pulmonary Hypertension group: n=25 patients with pulmonary hypertension (definition: pulmonary arterial pressure (PAP) above 25 mmHg)
- Valvular heart disease group: n=25 patients with valvular heart disease (at least moderate)
- Ischemic cardiomyopathy group: n=25 patients with ischemic cardiomyopathy
- HFpEF group: n=25 patients with HFpEF (heart failure with preserved ejection fraction, definition: EF over 50%, heart failure symptoms, elevated NT-proBNP over 400pg/ml)

SUMMARY:
BOLD measured with MRI may be a useful noninvasive method for the assessment of right ventricular O2 saturation. A validation of this method against right heart catheterization has not been fully performed. Whether the method may have a diagnostic and prognostic role in chronic heart failure patients is unclear.

DETAILED DESCRIPTION:
Measurement of blood oxygen saturation (O2 saturation) is essential for the clinical evaluation of patients with cardiovascular disease, heart failure, and pulmonary disease. With the introduction of the right heart catheter, measurements of O2 saturation in the right heart, venae cavae, and pulmonary artery became readily available and have thus contributed significantly to our hemodynamic understanding of congenital and acquired heart disease. Furthermore, the introduction of a pulmonary artery catheter, which can be implanted within minutes at the bedside, allows better monitoring for critically ill patients in the intensive care unit. In acquired heart disease, O2 saturation provides important information about systemic oxygen delivery and consumption, making it essential for evaluating heart failure patients and patients with pulmonary arterial hypertension. Nevertheless, invasive catheter implantation is associated with not insignificant risks of complications and a noninvasive method has not yet been established.

The blood oxygen level-dependent (BOLD) effect has been established in recent years as an effective method to noninvasively measure O2 saturation using T2 magnetic resonance imaging (T2-MRI). BOLD effect-based oximetry has been found to provide noninvasive information about both blood oxygenation, myocardial oxygenation, and skeletal muscle oxygenation using MRI. The principle underlying this technique exploits the dependence of the T2- relaxation time on the oxygenation of hemoglobin, as well as the different magnetic properties of hemoglobin in the oxygenated and deoxygenated states. To establish the mathematical relationship between the T2 relaxation time of whole blood and O2 saturation, a Luz-Meiboom (L-M) model describing the transverse (T2) relaxation arising from the transfer of protons between a protein and a water solution was proposed. The application of this model has improved the "classical" BOLD sequences, which were only measurable in static tissue (myocardium), minimizing the large estimation variability in flows (ventricles and vessels), allowing a more quantitative measurement. With the increasing number of patients receiving transcatheter aortic valve implantation (TAVI) as well as being diagnosed with atypical pulmonary hypertension, a large number of patients with relevant comorbidities require invasive hemodynamic evaluation. Simultaneous evaluation of central venous SO2 (ScvO2) and cardiac function is highly desirable and could allow noninvasive staging of frail high-risk patients. The first pilot clinical study of this concept was recently published.

The first aim of the investigators is to determine the precision of non-invasive O2 saturation measurement using BOLD-T2-MRI in contrast to invasive O2 saturation measurement using a right heart catheter in patients.

The secondary objective of the study is to investigate the role of BOLD measurements as a diagnostic test in patients with dyspnea at presentation, at least NYHA class 2 and an indication for cardio MRI. In these patients, BOLD measurements will be performed both at rest and during exercise. A sensitivity analysis will be performed to determine the diagnostic value of BOLD measurements in different patient populations.

ELIGIBILITY:
Inclusion Criteria:

Age > 18 years Ability to follow the study according to study protocol General ability to consent Presence of a written consent of the study participant Patients with a clinical indication for right heart catheterization

Exclusion Criteria:

Age <18 years. Pregnancy (for women of childbearing age, a pregnancy test is performed if pregnancy is possible) or breastfeeding.

Any condition that interferes with informed decision making General MRI exclusion criteria (pacemaker, defibrillator, intracranial aneurysm clips, metallic foreign bodies in the eyes) Any MRI exclusion criteria not listed here as determined by the performing MRI laboratory.

Hemodynamically unstable patients (heart rate < 50/min, systolic blood pressure < 90 mmHg, circulatory support devices: IABP, Impella) Complex supra- or ventricular arrhythmia occurring at rest or on exertion Right ventricular thrombus Recent pulmonary embolism Pulmonary instability (oxygen depletion or peripheral oxygen saturation <90%) Chronic lung disease (FEV< 35% on spirometry) Claustrophobia Sensorineural hearing loss from 30 dB and tinnitus

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All male and female patients (age ≥ 18 years) of the Cardiology Clinic at Campus Virchow Klinikum and Deutsches Herzzentrum Berlin will be screened with regard to inclusion and exclusion criteria. Patients eligible on the basis of these criteria will be included in the study after informed consent and written consent.
  I Part (validation) In the first part of the study (the validation), a total of 25 patients were to be scheduled for right heart catheterization.
  II part (clinical study) In the second part will be a total of 100 patients with dyspnea and clinical indication for MRI and 25 healthy control patients.
Sampling Method: Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
oxygenation within the blood measured with MRI versus catherization | 1 Year
  Comparison of the accuracy of BOLD MRI versus right heart catheterization (RHC)
differences in oxygenation within different heart failure groups | 1 Year
  Analysis of the sensitivity of BOLD measurements as a new diagnostic method for dyspnea at first presentation for various clinical applications

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Kelle, Principal Investigator — German Heart Center Berlin
Locations (1):
- Deutsches Herzzentrum Berlin, Berlin, Germany

REFERENCES:
- [Derived] Alogna A, Faragli A, Kolp C, Doeblin P, Tanacli R, Confortola G, Oetvoes J, Perna S, Stehning C, Nagel E, Pieske BM, Post H, Kelle S. Blood-Oxygen-Level Dependent (BOLD) T2-Mapping Reflects Invasively Measured Central Venous Oxygen Saturation in Cardiovascular Patients. JACC Cardiovasc Imaging. 2023 Feb;16(2):251-253. doi: 10.1016/j.jcmg.2022.08.020. Epub 2022 Nov 16. No abstract available. PMID 36648039